CLINICAL TRIAL: NCT02050607
Title: Fecal Microbiota Transplantation for the Treatment of Metabolic Syndrome
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Giovanni Cammarota, Prof, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMTandMETs-001; FMTandMETs-002 (Other: Catholic University of Sacred Heart - Rome)
Record Dates: First submitted 2013-11-07; First posted 2014-01-31 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Control group
- Fecal microbiota transplantation (Experimental): Fecal microbiota transplantation from healthy lean donors
  Interventions: Other: fecal microbiota transplantation from healthy lean donors

INTERVENTIONS:
Other: fecal microbiota transplantation from healthy lean donors — fecal microbiota transplantation from healthy lean donors
  Arms: Fecal microbiota transplantation

SUMMARY:
Obesity is associated with changes in the composition and metabolic function of the gut microbiota. Fecal microbiota transplantation (FMT), also known as "fecal bacteriotherapy" or "fecal infusion", refers to the process of injecting a liquid suspension of stool from a healthy donor into the gastrointestinal (GI) tract of a patient to cure a specific disease. However, since the recently established concept of human gut microbiome and its significant role in health and disease has caught on in the medical scientific world, this procedure has gained a great pathophysiological strength, meaning not only the simple infusion of stools, but the transplantation of a healthy gut microbiota in a patient with a disrupted one. In a recent dutch experience, FMT from lean donors was able to increase the insulin sensitivity in patients with metabolic syndrome.

Our primary aim is to evaluate if FMT from lean healthy donors, in association to lifestyle changes, is able to reduce insulin-resistance more than lifestyle changes alone in patients with metabolic syndrome.

All the patients with metabolic syndrome will receive lifestyle counselling (1400 kilocalories diet and physical activity encouragement), than will be randomized to FMT from healthy lean donors by upper endoscopy (group A) or no treatment (group B)

ELIGIBILITY:
Inclusion Criteria:

* Both males and females between 30 and 60 years old
* BMI>30 and >35 kg/m2
* Diagnosis of Metabolic Syndrome according to National Cholesterol Education Program's Adult Treatment Panel III criteria
* No ongoing therapy for diabetes, hyperlipidemia or arterial hypertension
* Signature of written informed consent

Exclusion Criteria:

* recent (3 months) use of probiotic, antibiotics or other drugs
* Increase in triglycerides levels, (≥ 300 mg/dl), LDL levels (≥ 190 mg/dl, or modification of body weight (±5%) during the last 3 months
* Relevant cardiovascular diseases or kidney diseases
* Relevant gastrointestinal diseases (such as inflammatory bowel disease or celiac disease)
* Former gastrointestinal surgery

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
difference in euglycemic clamp value at baseline and after the treatment | 6 months

SECONDARY OUTCOMES:
Disappearance of metabolic syndrome | 6 months
Modification in fasting blood glucose | 6 months
Modification in serum triglycerides | 6 months
Modification in serum High Density Lipoprotein cholesterol | 6 months
Modification in blood pressure | 6 months
Modification in abdominal circumference | 6 months
Modification in serum Tumor Necrosis Factor-alpha | 6 months
Modification in serum C-Reactive Protein | 6 months
Modification in serum interleukin-6 | 6 months
Modification in flow-mediated dilatation (FMD) of the brachial artery | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Sacred Heart - "A. Gemelli" University Hospital, Rome, Italy